CLINICAL TRIAL: NCT01104883
Title: The Efficacy of Adductor-Canal-Blockade on Morphine Consumption, Pain and Mobilisation After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Pia Jaeger MD, Department of Anaesthesia, Centre of Head and Orthopaedics, Rigshospitalet, Copenhagen, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-PJ-2009; 2009-017794-37 (EudraCT Number)
Record Dates: First submitted 2010-04-12; First posted 2010-04-16 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Total Knee Arthroplasty
Keywords: Adductor-Canal-Blockade; postoperative pain; US-guided nerve block; total knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adductor-Canal-Blockade (Experimental): Adductor-Canal-Blockade with ropivacaine
  Interventions: Procedure: Adductor-Canal-Blockade
- Adductor-Canal-blockade with saline (Placebo Comparator): Adductor-Canal-blockade with isotonic saline
  Interventions: Procedure: Adductor-Canal-blockade with saline

INTERVENTIONS:
Procedure: Adductor-Canal-Blockade — US-guided Adductor-Canal-Blockade with ropivacaine 7,5 mg/ml
  Other Names: Naropine; Postoperative pain; US-guided nerve block
  Arms: Adductor-Canal-Blockade
Procedure: Adductor-Canal-blockade with saline — US-guided Adductor-Canal-blockade with saline
  Other Names: placebo block
  Arms: Adductor-Canal-blockade with saline

SUMMARY:
The purpose of this study is to determine whether Adductor-Canal-Blockade is effective at reducing morphine consumption and pain, and at the same time improving mobilisation after total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Total Knee Arthroplasty in spinal anaesthesia
* ASA 1-3
* BMI 18-40
* Written informed consent

Exclusion Criteria:

* Can not cooperate to the exam
* Do not speak or understand Danish
* Drug allergy
* Alcohol or drug abuse
* Daily consumption of strong opioids
* Unable to complete the Timed Up and Go test preoperatively

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 0-24 hours postoperative
  Total morphine consumption at the interval 0-24 hours postoperative.

SECONDARY OUTCOMES:
Total morphine consumption | 0-26 hours postoperative
  Total morphine consumption at the intervals 0-2, 0-4, 0-8 and 0-26 hours postoperative.
Pain during rest | 0-26 hours postoperative
  0-100 mm at a visual analogue scale (VAS), at the intervals 2, 4, 8, 24 and 26 hours postoperative, and the area under the curve for the intervals 2-24 and 24-26 hours postoperative.
Pain during 45 degrees active flexion of the knee | 0-26 hours postoperative
  0-100 mm at a visual analogue scale (VAS), at the intervals 2, 4, 8, 24 and 26 hours postoperative, and the area under the curve for the intervals 2-24 and 24-26 hours postoperative.
A change in pain in the placebo group | 24-26 hours postoperative
  0-100 mm at a visual analogue scale (VAS), at the intervals 24 and 26 hours postoperative.
Postoperative nausea | 0-26 hours postoperative
  Nausea scores(0-3)at 2,4,8,24,26 hours postoperative.
Zofran consumption | 0-26 hours postoperative
  Total zofran consumption at the intervals 0-24 and 24-26 hours postoperative.
Sedation | 0-26 hours postoperative
  Seadtion score (0-3) at 2,4,8,24,26 hours postoperative.
Mobilisation | 20-26 hours postoperative
  Number of seconds it takes to complete the "Timed Up and Go" test, at 20 and 26 hours postoperative.
Postoperative vomiting | 0-26 hours postoperative
  Number of vomiting episodes at the intervals 0-2,2-4,4-8,8-24,24-26 hours postoperative.

CONTACTS AND LOCATIONS:
Overall Officials: Pia Jæger, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Department of Anaesthesia, Privathospitalet Hamlet, Frederiksberg, Denmark, Copenhagen, Frederiksberg
  - Department of Surgery and Anaesthesia, Glostrup Hospital, Glostrup Municipality, Glostrup

REFERENCES:
- [Derived] Jenstrup MT, Jaeger P, Lund J, Fomsgaard JS, Bache S, Mathiesen O, Larsen TK, Dahl JB. Effects of adductor-canal-blockade on pain and ambulation after total knee arthroplasty: a randomized study. Acta Anaesthesiol Scand. 2012 Mar;56(3):357-64. doi: 10.1111/j.1399-6576.2011.02621.x. Epub 2012 Jan 4. PMID 22221014